

## **COVER SHEET**

Date: 7/12/2017

**VALIDATION PROTOCOL #276** 

Title: Plan for Testing Fingerstick bloods on Magellan Systems

Sponsor:

Magellan Diagnostics

101 Billerica Ave.,

North Billerica, Ma. 01862

Reba Daoust Director of QA/RA 978-248-4811

Investigator: Peter Rappo, MD

Pediatrician

Pediatric Associates, Inc. 370 Oak St., Suite A Brockton, Ma. 02301 Phone: 508-584-1210

- 3 Sites total for Dr. Peter Rappo
- Site Registration forms submitted

Approved

JUL 21 2017

Aspire IRB

Received

JUL 1 7 2017

Aspire IRB